CLINICAL TRIAL: NCT06897787
Title: The Effect Of Different Proximal Segment Positioning Methods On Postoperative Condylar Remodeling in Patients Undergoing Bimaxillary Orthognathic Surgery
Brief Title: Effect of Proximal Segment Positioning on Postoperative Condylar Remodeling in Bimaxillary Orthognathic Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07.03.2025-E.185561
Record Dates: First submitted 2025-03-17; First posted 2025-03-27 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dentofacial Deformities; Dentofacial Anomalies [Including Malocclusion] and Other Disorders of Jaw (M26-M27)
Keywords: mandibular condyle; orthognathic surgery; manuel condyle positioning
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: Manuel positioning group (Active Comparator): This is the group in which leveling between the lower border of the proximal segment and the mandibular base is achieved through proximal segment rotation after mandibular osteotomies.
  Interventions: Procedure: manuel positioning group
- group 2: mandibular basis osteotomy (Experimental): This is the group in which the proximal segment is left in its preoperative position, and leveling of the mandibular base is achieved by performing an osteotomy on the lower border of the proximal segment.
  Interventions: Procedure: mandibular basis osteotomy

INTERVENTIONS:
Procedure: manuel positioning group — As Prof. Reyneke does, mandibular base and proximal segment leveling are performed first, followed by fixation.
  Arms: group 1: Manuel positioning group
Procedure: mandibular basis osteotomy — After the mandibular sagittal split, secure the proximal segment in its preoperative position and remove the bone piece for leveling. After that, fixation is performed.
  Arms: group 2: mandibular basis osteotomy

SUMMARY:
Bimaxillary orthognathic surgery is a surgical procedure that involves simultaneous corrections to both the maxilla (upper jaw) and mandible (lower jaw). This surgery is performed to correct facial and jaw deformities, improve occlusion, and enhance facial symmetry. The need for orthognathic surgery typically arises in cases where there is a significant discrepancy between the upper and lower jaws or severe malocclusion.

In bimaxillary orthognathic surgery, following mandibular osteotomies, the lower jaw is divided into two segments: the distal segment, which contains the teeth, and the proximal segment, which includes the condylar head. While the distal segment is positioned according to the ideal occlusion planned in collaboration with orthodontists using digital design, the management of the proximal segment varies among surgeons. Some surgeons leave the proximal segment in its original position without mobilization, whereas others reposition it through rotational movements.

This study aims to evaluate condylar remodeling by comparing these two surgical approaches in patients divided into two groups, assessing how each technique affects postoperative outcomes.

DETAILED DESCRIPTION:
Bimaxillary orthognathic surgery is a surgical procedure that involves simultaneous correction of both the maxilla (upper jaw) and the mandible (lower jaw). This surgery is performed to correct facial and jaw deformities, improve occlusion, and enhance facial symmetry. The need for orthognathic surgery typically arises in cases where there is a discrepancy between the upper and lower jaws or significant malocclusion.

In bimaxillary orthognathic surgery, following mandibular osteotomies, the lower jaw is divided into two segments: the distal segment, which contains the teeth, and the proximal segment, which includes the condylar head. While the distal segment is positioned according to the ideal occlusion planned in collaboration with orthodontists using digital design, the management of the proximal segment varies among surgeons. Some surgeons leave the proximal segment in its original position without mobilization, whereas others reposition it through rotational movements.

This study aims to evaluate condylar remodeling by applying both surgical approaches to patients divided into two groups. The study will assess how each surgical technique affects condylar remodeling both in terms of angular and volumetric changes, determining which approach better preserves and reshapes the joint optimally. Ultimately, the findings will contribute to the future course of bimaxillary orthognathic surgeries and their benefits for patients.

Since 1990, cone-beam computed tomography (CBCT) has been effectively used in oral and maxillofacial surgery as an alternative to conventional computed tomography (CT). Compared to CT, CBCT has demonstrated advantages such as requiring a lower radiation dose, producing fewer metal artifacts, being more accessible, and offering easier usage. Due to these advantages, CBCT has been successfully utilized in oral implant applications, where a localized focus area is necessary. However, limitations such as low contrast range, restricted detector size, limited soft tissue information, increased noise due to scattered radiation, and a subsequent loss of contrast resolution, along with its inability to determine Hounsfield units (HU), restrict its use in maxillofacial applications.

Particularly in preoperative digital planning for orthognathic surgery and subsequent evaluations, it is crucial to select an appropriate HU range to segment the maxilla and mandible and accurately transfer all topographic features into the digital domain. This step forms the foundation of patient-specific virtual surgical planning, which requires the use of computed tomography (CT) for optimal execution. Studies have preferred CT as the imaging method due to its high accuracy in topographic transfer and its ability to provide precise cortical bone thickness, a critical factor for designing patient-specific guides and plates. For these reasons, we also plan to use CT imaging in our study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients planned to undergo bimaxillary orthognathic surgery with Class III skeletal deformity
2. Patients aged 18-65
3. Patients who have undergone preoperative orthodontic treatment
4. Patients who, after mandibular distal segment sagittal split osteotomy, exhibit a maximum of 4 degrees of counterclockwise rotation when brought to the final position

Exclusion Criteria:

1. Patients with a history of joint surgery, orthognathic surgery, or tumor resection
2. Patients with facial asymmetry
3. Patients with cleft lip and palate syndrome, craniofacial syndrome, or trauma
4. Patients who, after mandibular distal segment sagittal split osteotomy, exhibit more than 4 degrees of counterclockwise rotation when brought to the final position (as the amount of base resection required in this case would exceed feasible limits).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
mandibular condyle position superimposition | 2 year
  During bimaxillary orthognathic surgery, proximal segment positioning devices will be used in both groups to ensure that the condylar position remains at the location determined during virtual surgical planning. These devices will be custom-designed for each patient by the researchers using the virtual surgical planning software and printed using an in-house 3D printer. These positioning devices will maintain the condyle in its initial position during mandibular fixation. Postoperative DICOM data obtained from computed tomography images will be used to superimpose the condylar positions, and the amount of displacement in three planes (x, y, z) will be measured in millimeters (mm). Additionally, condylar volume changes will be calculated in cubic centimeters (cm³) using the superimposition method, and differences between the groups will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided